CLINICAL TRIAL: NCT02530242
Title: Point-of-Care End-Tidal Carbon Monoxide Measurement to Screen for Sickle Cell Disease
Brief Title: Carbon Monoxide Measurement to Screen for Sickle Cell Disease
Acronym: SCDCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Capnia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-013
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- End-tidal Carbon Monoxide Subjects (Other): Children between 1-18 years old with Sickle Cell Anemia
  Interventions: Device: End-tidal Carbon Monoxide Subjects
- End-tidal Carbon Monoxide Controls (Other): Healthy children age matched with subjects.
  Interventions: Device: End-tidal Carbon Monoxide Controls

INTERVENTIONS:
Device: End-tidal Carbon Monoxide Subjects — ETCO monitor will be used to measure CO levels in subjects and controls.
  Arms: End-tidal Carbon Monoxide Subjects
Device: End-tidal Carbon Monoxide Controls — ETCO monitor will be used to measure CO levels in subjects and controls.
  Arms: End-tidal Carbon Monoxide Controls

SUMMARY:
Modify the design of the CoSense device (Model C20112, currently cleared by the FDA for ETCO (end-tidal carbon monoxide) monitoring to improve accuracy and consistency under temperature conditions encountered in countries with high prevalence of SCD (Sickle Cell Disease).

DETAILED DESCRIPTION:
Increase the temperature operating range of ETCO measurements to 5 to 45°C. The signal output-to-CO (carbon monoxide) concentration correlation of the CO sensor is dependent on temperature. The new algorithm will be a different approach because the current algorithm is at the limits of its capability. We will establish the new specifications by determining performance in a bench model under simulated temperature conditions. We will then determine the ability of the modified device to distinguish between SCD and healthy controls. During this initial testing, we will examine the validity of ETCO measurements under regulated room temperature in the hospital setting. We will enroll 20 subjects, 10 each in the SCD arm and control arm to determine the mean and variance of the ETCO values.

ELIGIBILITY:
Inclusion Criteria:

* Parental / legal guardian consent
* Subject assent for participants ages 7 and above
* Male and female children ages 1-18 years old
* For Hb SS (Homozygous sickle cell anemia) subjects, hemoglobin baseline hemoglobin ≤10 g/dL based upon average hemoglobin value in past year

Exclusion Criteria:

* Subjects must not meet any of the following exclusion criteria to be considered eligible for study enrollment:
* Had a red blood cell transfusion within 8 weeks prior to enrollment
* Currently a primary smoker or was a primary smoker within 4 weeks prior to enrollment
* Exposed to second hand smoke within 24 hours prior to breath sample collections
* Have current upper respiratory infection or symptomatic asthma
* For healthy subjects, known to have the sickle cell trait by electrophoresis or genetic testing

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Lal, MD, Principal Investigator — Children's Hospital & Research Center at Oakland

REFERENCES:
- [Background] Lal A, Patterson L, Goldrich A, Marsh A. Point-of-care end-tidal carbon monoxide reflects severity of hemolysis in sickle cell anemia. Pediatr Blood Cancer. 2015 May;62(5):912-4. doi: 10.1002/pbc.25447. Epub 2015 Feb 14. PMID 25683629

RESULTS

PARTICIPANT FLOW:
Groups:
- End-tidal Carbon Monoxide Controls: Healthy children age and gender matched with subjects.
  End-tidal Carbon Monoxide Controls: ETCO monitor will be used to measure CO levels in subjects and controls.
Period: Overall Study
Arm/Group | End-tidal Carbon Monoxide Subjects | End-tidal Carbon Monoxide Controls
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — excluded due to asthma and oxcarbazepine | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | End-tidal Carbon Monoxide Subjects | End-tidal Carbon Monoxide Controls | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Full Range); unit: years] | 9.4 [5 to 14] | 9.7 [5 to 14] | 9.5 [5 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: End-Tidal Carbon Monoxide
Description: Compare ETCO between subjects and controls
Time Frame: 1 hour
Measure: Median (Full Range); unit: ppm
Arm/Group | End-tidal Carbon Monoxide Subjects | End-tidal Carbon Monoxide Controls
Number analyzed (Participants) | 16 | 15
ppm | 4.35 [1.8 to 9.7] | .80 [.2 to 2.3]

ADVERSE EVENTS:
Arm/Group | End-tidal Carbon Monoxide Subjects | End-tidal Carbon Monoxide Controls
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
A limitation of the data is the small number of subjects and that it was conducted under controlled circumstances in the clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes